CLINICAL TRIAL: NCT02174991
Title: A Prospective Study to Assess the Hypotensive Efficacy of Rho-Kinase Inhibitor AR-12286 Ophthalmic Solution 0.5% and 0.7% in Glaucoma Patients With Uncontrolled Intraocular Pressure to Avoid Surgical Intervention
Brief Title: A Compassionate Case Study to Assess the Hypotensive Efficacy of Rho-Kinase Inhibitor AR-12286 Ophthalmic Solution 0.5% and 0.7% in Glaucoma Patients With Uncontrolled Intraocular Pressure to Avoid Surgical Intervention
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York Glaucoma Research Institute (Other)
Responsible Party: Principal Investigator, Jessica Jasien, Co-Investigator, New York Glaucoma Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14.15
Record Dates: First submitted 2014-06-17; First posted 2014-06-26 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — AR-12286

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 0.5% Rho-Kinase Inhibitor (Experimental): AR-12286 is a novel Rho-kinase inhibitor developed by Aerie Pharmaceuticals, Inc., Bridgewater, NJ. It is a potent Rho-kinase inhibitor with single-digit nanomolar inhibitory activity against Rho-kinase in enzymatic inhibition assays (deLong MA, et al. IOVS 2009; 50: ARVO E-abstract 4058). Mechanism-of action studies in monkeys demonstrate that AR-12286 lowers IOP primarily by increasing aqueous humor outflow through the trabecular meshwork (Wang RF, et al. IOVS 2009; 50:ARVO E-abstract 1465). Rho-kinase AR-12286 is well tolerated and produces clinically and statistically significant ocular hypotensive efficacy in patients with ocular hypertension and glaucoma. It is well tolerated by most of patients and the only side effect was ocular hyperemia in a minority of subjects (Williams, Novack, Van Haarlem, & Kopczynski, 2011). It is currently in phase II testing.
  Interventions: Drug: Rho-Kinase Inhibitor (AR-12286)
- 0.7% Rho-Kinase Inhibitor (Experimental): AR-12286 is a novel Rho-kinase inhibitor developed by Aerie Pharmaceuticals, Inc., Bridgewater, NJ. It is a potent Rho-kinase inhibitor with single-digit nanomolar inhibitory activity against Rho-kinase in enzymatic inhibition assays (deLong MA, et al. IOVS 2009; 50: ARVO E-abstract 4058). Mechanism-of action studies in monkeys demonstrate that AR-12286 lowers IOP primarily by increasing aqueous humor outflow through the trabecular meshwork (Wang RF, et al. IOVS 2009; 50:ARVO E-abstract 1465). Rho-kinase AR-12286 is well tolerated and produces clinically and statistically significant ocular hypotensive efficacy in patients with ocular hypertension and glaucoma. It is well tolerated by most of patients and the only side effect was ocular hyperemia in a minority of subjects (Williams, Novack, Van Haarlem, & Kopczynski, 2011). It is currently in phase II testing.
  Interventions: Drug: Rho-Kinase Inhibitor (AR-12286)

INTERVENTIONS:
Drug: Rho-Kinase Inhibitor (AR-12286)

SUMMARY:
A. To evaluate the ocular hypotensive efficacy of the rho-kinase Inhibitor (AR-12286 0.5% and 0.7%) ophthalmic solutions in open-angle glaucoma patients with uncontrolled IOP who are facing surgical intervention. Patients will be treated for 6 months in this initial trial.

B. To evaluate the efficacy of AR-12286 in enabling treated patients to delay or avoid the necessity of surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with open-angle glaucoma.
2. IOP above the target range or visual field progression with use of maximum standard drug therapy.
3. Have given written informed consent, prior to any investigational procedures.
4. Ability to attend for the 6-month duration of treatment.

Exclusion Criteria:

1. Angle-closure glaucoma
2. Eyes having had previous incisional glaucoma surgery
3. Known hypersensitivity to any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics.
4. Ocular medication of any kind within 30 days of base-line visit, with the exception of ocular hypotensive medications and/or lubricating drops for dry eye (which may be used throughout the study).
5. Any abnormality preventing reliable applanation tonometry of the treated eye.
6. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
7. Participation in any investigational study within the past 30 days.
8. Inability to perform reliable visual field testing.
9. Unwilling to sign the consent form approved by the Institutional Review Board (IRB) of the New York Eye and Ear Infirmary.
10. Self-reported poor compliance to treatment.
11. Reluctance to return for scheduled follow-up visits.
12. Patients not able to understand the nature of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
IOP Reduction | 6 Months
  Avoid surgical intervention of glaucoma treatment with use of AR-12286; long lasting effect of study drug to reduce IOP by increase of aqueous outflow

SECONDARY OUTCOMES:
Tolerance and Lasting IOP Effect | 6 Months
  To evaluate the ocular hypotensive safety (tolerance) of Rho-Kinase Inhibitor (AR-12286 0.5% and 0.7%) ophthalmic solution in patients who are avoiding surgical intervention and the long last effect of IOP reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Glaucoma Associates of New York, New York, New York, United States